CLINICAL TRIAL: NCT02046408
Title: Computer-Facilitated 5A's for Smoking Cessation in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01DA034253-01 (NIH)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Nicotine Addiction; Smoking Cessation
Keywords: Smoking; 5A's for smoking cessation; tailored health messages; Patient-facing information technology; Mobile health; behavioral health
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet Intervention (Experimental): Primary care providers will be randomized into intervention or control conditions. The patients of intervention providers will be given a computer tablet that provides 5A's for smoking cessation counseling. Patients of control providers will not receive a tablet intervention.
  Interventions: Other: Computer Tablet
- Control (No Intervention): Primary care providers will be randomized into intervention or control conditions. The patients of intervention providers will be given a computer tablet that provides 5A's for smoking cessation counseling. Patients of control providers will not receive a tablet intervention.

INTERVENTIONS:
Other: Computer Tablet
  Arms: Tablet Intervention

SUMMARY:
This study tests the use of handheld computer tablets to promote the integration of 5A's (Ask, Advise, Assess, Assist, Arrange) for smoking cessation in academic and community primary care clinics. Although most patients receive the "ask" and "advise" steps, only slightly more than half are "assessed" for readiness to change, less than half receive "assistance" in changing, and only 9% have an "arranged" follow-up. While the large majority of primary care providers support the 5A's model, negative attitudes and the lack of time, knowledge, and cessation skills are common obstacles. Alternate service delivery systems that address these obstacles and evidence-based strategies to promote their implementation are needed to improve provider adherence and 5A's fidelity.

DETAILED DESCRIPTION:
This project develops and tests a computer-facilitated 5A's (CF-5A's) model that administers the 5A's intervention to patients then prompts providers for reinforcing next steps. CF-5A's could efficiently and effectively promote smoking cessation while educating providers about cessation resources and appropriate follow-up. Based on the Technology Acceptance Model, clinically tailored strategies to promote CF-5A's implementation will be developed and tested to ensure the appropriate use and uptake of this new service delivery model. Development of the model, materials, and strategies will occur in years 1 and 2.

Baseline data collection occurs in year 2, followed by a randomized trial of CF- 5A's where the provider is the unit of randomization. Provider use of the 5A's will primarily be assessed with a brief phone call to the patient after the primary care visit has occurred.

Although focused on 5A's for smoking cessation, this study examines the underlying implementation science of computer-aided service delivery models with important implications for the integration of other substance use or behavioral health interventions in primary care. Implementation factors will be assessed using qualitative interviews and brief pre-post surveys.

ELIGIBILITY:
Inclusion Criteria: All primary care providers and clinic staff are eligible to participate. Patients must have

* a primary care appointment
* smoked a cigarette in past 7 days
* smoked at least 100 cigarettes in lifetime
* speak English or Spanish
* be cognitively able to use computer tablet

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Does not speak English or Spanish
* acute intoxication on alcohol or illicit drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
5A's Fidelity | Baseline assessment 2013-14; Intervention 2014-2015
  Baseline and post-tablet intervention assessments of primary care provider adherence to 5A's protocol for smoking cessation. Patients are called after their primary care appointment and asked a series of questions to determine if (and which of) the 5A's were used during that visit.

SECONDARY OUTCOMES:
Tablet Usage | 7/2014-7/2015
  Intervention includes system strategies to improve usage of computer tablets in primary care waiting rooms. Outcome = tablet saturation or proportion of patients given a tablet.

OTHER OUTCOMES:
Implementation Factors | July 2013-2015
  Qualitative interview data to assess the utility of the "Technology Acceptance Model" in explaining tablet and 5A's usage. Variables assessed include perceived usefulness, social norms and influence, and facilitating conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Satterfield, PhD, Principal Investigator — University of California
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - UCSF Adult Primary Care Mt. Zion Clinic, San Francisco, California

REFERENCES:
- [Derived] Satterfield JM, Gregorich SE, Kalkhoran S, Lum PJ, Bloome J, Alvarado N, Munoz RF, Vijayaraghavan M. Computer-Facilitated 5A's for Smoking Cessation: A Randomized Trial of Technology to Promote Provider Adherence. Am J Prev Med. 2018 Jul;55(1):35-43. doi: 10.1016/j.amepre.2018.04.009. Epub 2018 Jun 18. PMID 29929682